CLINICAL TRIAL: NCT02799745
Title: A Randomized Study of Enzalutamide in Patients With Localized Prostate Cancer Undergoing Active Surveillance (ENACT)
Brief Title: A Randomized Study of Enzalutamide in Patients With Localized Prostate Cancer Undergoing Active Surveillance
Acronym: ENACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9785-MA-1010
Record Dates: First submitted 2016-02-29; First posted 2016-06-15 (Estimated); Results first posted 2021-11-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Therapeutic Cancer Progression; Pathological Cancer Progression; Enzalutamide; Prostate Cancer; Active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enzalutamide (Active Comparator): Participants received 160-milligrams (mg) enzalutamide administered as four 40-mg capsules, orally once daily for 1 year of treatment period. Following the 1-year treatment period, all participants were followed for 1 additional year. Post the 1-year follow-up period, participants then started the continued follow-up period, in which, participants were followed up every 3 months for these 2 years, after which follow-up was either every 6 months up to 36 months or until the end of study (total duration of follow up in the study was approximately up to 35.9 months).
  Interventions: Drug: Enzalutamide
- Active Surveillance (AS) (Other): Participants did not receive any study treatment in this arm but were on continued active surveillance (AS) for 1 year of treatment period. Following the 1-year treatment period, all participants were followed for 1 additional year. Post the 1-year follow up, participants then started the continued follow-up period, in which, participants were followed up every 3 months for these 2 years, after which follow-up was either every 6 months up to 36 months or until the end of study (total duration of follow up in the study was approximately up to 35.9 months).
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide
Other: Active Surveillance
  Arms: Active Surveillance (AS)

SUMMARY:
The primary purpose of this study was to compare the time to prostate cancer progression (pathological or therapeutic progression) between patients treated with enzalutamide versus patients undergoing active surveillance.

DETAILED DESCRIPTION:
This was a multicenter, randomized, open label exploratory study, conducted in the US and Canada, evaluating the efficacy and safety of enzalutamide for extension of time to prostate cancer progression (pathological or therapeutic) in patients with clinically localized, histologically proven prostate cancer that is categorized as low risk or intermediate risk and who were under AS.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate diagnosed (with ≥10 core biopsy) within 6 months of screening. The biopsy that was used for this diagnosis must be submitted for central pathology review.
* Prostate cancer categorized (as determined by central pathology review) as low risk is defined as T1c-T2a, PSA<10, N0, M0 (or presumed N0, M0 if CT/bone scan not done due to low risk of metastases), GS ≤ 6, ECOG status ≤2 and estimated life expectancy >5 years OR intermediate risk is defined as T2b-T2c, PSA<20, N0, M0 (or presumed N0, M0 if CT/bone scan not done), GS ≤7 (3+4 pattern only), ECOG status ≤ 2 and estimated life expectancy > 5 years. Prostate cancer categorized (as determined by central pathology review) to the very low risk category (T1c, GS ≤6, PSA <10 ng/mL, fewer than 3 prostate biopsy cores positive,

  ≤50% cancer in any core, PSA density <0.15 ng/mL/g) is not included.
* Ability to swallow study drugs and to comply with study requirements throughout the study
* Institutional Review Board (IRB)-/Independent Ethics Committee (IEC)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures
* Throughout study, male subject and a female partner who is of childbearing potential must use two acceptable methods of birth control (one of which must include a condom barrier method of contraception) starting at screening and continuing throughout the study period and for three months after the final study drug administration. Two acceptable methods of birth control thus include the following:

  1. Condom (barrier method of contraception) AND
  2. One of the following is required:

  i. Established use of oral, injected or implanted hormonal methods of contraception by the female partner; ii. Placement of an intrauterine device or intrauterine system by the female partner; iii. Additional barrier method: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam / gel / film / cream / suppository by the female partner; iv. Tubal ligation in the female partner.
* Must not donate sperm starting at screening throughout the study period and for 90 days after the final study drug administration.

Exclusion Criteria:

* Prior radiotherapy, surgery, chemotherapy, or hormonal therapy for prostate cancer
* Very low risk category (T1c, GS ≤6, PSA <10 ng/mL, fewer than 3 prostate biopsy cores positive, ≤50% cancer in any core, PSA density <0.15 ng/mL/g)
* Prior transurethral resection of the prostate or prior transurethral microwave thermotherapy of the prostate
* Use of oral glucocorticoids within 1 month of screening
* Use of 5 alpha reductase inhibitor within 1 month of screening or total use, within the last two years prior to screening, of >3 months
* Presence of metastatic disease
* History of seizure or any condition that may predispose to seizures at any time in the past. History of loss of consciousness or transient ischemic attack within 12 months of screening
* Absolute neutrophil count < 1,500/μL, platelet count < 100,000/μL, or hemoglobin < 6.2 mmol/L (10 g/dL) at screening
* Total bilirubin >1.5 times the upper limit of normal (ULN) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 X ULN at screening
* Creatinine > 177 μmol/L (> 2 mg/dL) at screening
* Albumin < 30 g/L (3.0 g/dL) at screening
* Major surgery within 4 weeks prior to Randomization Visit
* Clinically significant cardiovascular disease including:

  1. Myocardial infarction or uncontrolled angina within 6 months
  2. Congestive heart failure New York Heart Association (NYHA) class 3 or 4
  3. History of clinically significant ventricular arrhythmias
  4. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  5. Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mm Hg) at screening
  6. Bradycardia as indicated by a heart rate of < 45 beats per minute on the screening electrocardiogram (ECG) and on physical examination
  7. Uncontrolled hypertension as indicated by at least 2 consecutive measurements of a resting systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening Visit
* Known hypersensitivity to enzalutamide or any of its components.
* Subject has received investigational therapy within 28 days or 5 half lives, whichever is longer, prior to screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (54):
- United States (50):
  - Site US10034, Birmingham, Alabama
  - Site US10024, Homewood, Alabama
  - Site US10007, Tucson, Arizona
  - Site US10055, Tucson, Arizona
  - Site US10004, Los Angeles, California
  - Site US10026, Sacramento, California
  - Site US10010, San Diego, California
  - Site US10051, Aurora, Colorado
  - Site US10029, Denver, Colorado
  - Site US10054, Denver, Colorado
  - Site US10072, Bradenton, Florida
  - Site US10057, Lakeland, Florida
  - Site US10038, Chicago, Illinois
  - Site US10062, Chicago, Illinois
  - Site US10074, Chicago, Illinois
  - Site US10018, Glenview, Illinois
  - Site US10071, Lake Barrington, Illinois
  - Site US10046, Carmel, Indiana
  - Site US10009, Jeffersonville, Indiana
  - Site US10037, New Orleans, Louisiana
  - Site US10006, Shreveport, Louisiana
  - Site US10001, Towson, Maryland
  - Site US10032, Boston, Massachusetts
  - Site US10008, Troy, Michigan
  - Site US10069, Lincoln, Nebraska
  - Site US10044, Omaha, Nebraska
  - Site US10067, Omaha, Nebraska
  - Site US10061, Lebanon, New Hampshire
  - Site US10049, Morristown, New Jersey
  - Site US10043, Voorhees Township, New Jersey
  - Site US10068, Brooklyn, New York
  - Site US10050, Cheektowaga, New York
  - Site US10030, Garden City, New York
  - Site US10028, Poughkeepsie, New York
  - Site US10021, Syracuse, New York
  - Site US10022, Syracuse, New York
  - Site US10047, Gastonia, North Carolina
  - Site US10045, Cleveland, Ohio
  - Site US10015, Middleburg Heights, Ohio
  - Site US10053, Oklahoma City, Oklahoma
  - Site US10063, Bala-Cynwyd, Pennsylvania
  - Site US10052, Lancaster, Pennsylvania
  - Site US10014, Warwick, Rhode Island
  - Site US10019, Myrtle Beach, South Carolina
  - Site US10011, Nashville, Tennessee
  - Site US10056, Dallas, Texas
  - Site US10036, Houston, Texas
  - Site US10035, San Antonio, Texas
  - Site US10058, Richmond, Virginia
  - Site US10017, Milwaukee, Wisconsin
- Canada (4):
  - Site CA15005, Abbotsford, British Columbia
  - Site CA15004, Halifax, Nova Scotia
  - Site CA15001, Toronto, Ontario
  - Site CA15003, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Handa N, Shore ND, Cooperberg MR, Davicioni E, Zhao X, Elsouda D, Liu Y, Proudfoot JA, Kuperman G, Russell D, Iwata KK, Schaeffer EM, Ross A. Transcriptome profiling of prostatic tumours from ENACT trial patients with or without enzalutamide. BJU Int. 2025 Nov;136(5):920-929. doi: 10.1111/bju.16861. Epub 2025 Jul 31. PMID 40742002
- [Derived] Ross AE, Iwata KK, Elsouda D, Hairston J, Russell D, Davicioni E, Proudfoot JA, Shore ND, Schaeffer EM. Transcriptome-Based Prognostic and Predictive Biomarker Analysis of ENACT: A Randomized Controlled Trial of Enzalutamide in Men Undergoing Active Surveillance. JCO Precis Oncol. 2024 Apr;8:e2300603. doi: 10.1200/PO.23.00603. PMID 38635932
- [Derived] Shore ND, Renzulli J, Fleshner NE, Hollowell CMP, Vourganti S, Silberstein J, Siddiqui R, Hairston J, Elsouda D, Russell D, Cooperberg MR, Tomlins SA. Enzalutamide Monotherapy vs Active Surveillance in Patients With Low-risk or Intermediate-risk Localized Prostate Cancer: The ENACT Randomized Clinical Trial. JAMA Oncol. 2022 Aug 1;8(8):1128-1136. doi: 10.1001/jamaoncol.2022.1641. PMID 35708696
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=9785-MA-1010
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14506&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with clinically localized, histologically proven prostate cancer diagnosed within 6 months of screening and had been on active surveillance were enrolled in this study. Participants were categorized as low risk or intermediate risk and had a minimum of 10 cores from transrectal ultrasound-guided prostate biopsy (multiparametric magnetic resonance imaging [mpMRI]-targeted versus non-mpMRI-targeted) done within 6 months prior to screening visit.
Pre-assignment Details: Randomization was stratified according to prostate cancer risk (low and intermediate) and type of biopsy performed (mpMRI-targeted and non-mpMRI-targeted). Out of 310 participants who were screened, 83 participants were considered screen failures.
Groups:
- Enzalutamide: The study has 3 parts: treatment period, 1 year follow-up period and continued follow-up period. Participants received 160-miligram (mg) enzalutamide administered as four 40-mg capsules, orally once daily for 1 year of treatment period. Following the 1-year treatment period, all participants were followed for 1 additional year. Post the 1-year follow-up period, participants then started the continued follow-up period, in which, participants were followed up every 3 months for these 2 years, after which follow-up was either every 6 months up to 36 months or until the end of study (total duration of follow up in the study was approximately up to 35.9 months).
- Active Surveillance: The study has 3 parts: treatment period, 1 year follow-up period and continued follow-up period. Participants did not receive any study treatment in this arm but were on continued active surveillance (AS) for 1 year of treatment period. Following the 1-year treatment period, all participants were followed for 1 additional year. Post the 1-year follow up, participants then started the continued follow-up period, in which, participants were followed up every 3 months for these 2 years, after which follow-up was either every 6 months up to 36 months or until the end of study (total duration of follow up in the study was approximately up to 35.9 months).
Period: Overall Study
Arm/Group | Enzalutamide | Active Surveillance
Started | 114 | 113
Treated | 112 | 113
Completed | 58 | 42
Not Completed | 56 | 71
Not completed — Participant moved out of state | 1 | 0
Not completed — Discontinued due to planned surgery | 1 | 0
Not completed — Withdrawal by Subject | 16 | 25
Not completed — Protocol Deviation | 4 | 5
Not completed — Progressive Disease | 28 | 38
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 3 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were randomized.
Groups:
- Enzalutamide: The study has 3 parts: treatment period, 1 year follow-up period and continued follow-up period. Participants received 160-mg enzalutamide administered as four 40-mg capsules, orally once daily for 1 year of treatment period. Following the 1-year treatment period, all participants were followed for 1 additional year. Post the 1-year follow-up period, participants then started the continued follow-up period, in which, participants were followed up every 3 months for these 2 years, after which follow-up was either every 6 months up to 36 months or until the end of study (total duration of follow up in the study was approximately up to 35.9 months).
- Active Surveillance: The study has 3 parts: treatment period, 1 year follow-up period and continued follow-up period. Participants did not receive any study treatment in this arm but were on continued AS for 1 year of treatment period. Following the 1-year treatment period, all participants were followed for 1 additional year. Post the 1-year follow up, participants then started the continued follow-up period, in which, participants were followed up every 3 months for these 2 years, after which follow-up was either every 6 months up to 36 months or until the end of study (total duration of follow up in the study was approximately up to 35.9 months).
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | Active Surveillance | Total
Number analyzed (Participants) | 114 | 113 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (8.18) | 66.9 (7.27) | 66.1 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 114 | 113 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 108 | 107 | 215
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 105 | 99 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Type of Biopsy [Count of Participants; unit: Participants] — Type of biopsies included: 1. mpMRI (multiparametric magnetic resonance imaging) type, 2. non-mpMRI type.
  Participants
    mpMRI-targeted | 27 | 28 | 55
    non-mpMRI-targeted | 87 | 85 | 172
Prostate Cancer Risk [Count of Participants; unit: Participants] — Low risk:no higher than T1c-T2a, prostate specific antigen(PSA)<10,N0,M0(or presumed N0,M0 if computerized tomography[CT]/bone scan not done due to low risk of metastases),gleason score(GS)<=6,eastern cooperative oncology group(ECOG)status<= 2, life expectancy>5years. Intermediate risk:no higher than T2b-T2c, PSA<20, N0, M0(or presumed N0, M0 if CT/bone scan not done), GS<=7(3+4 pattern only),ECOG status<=2, life expectancy>5 years. No primary GS 4 was allowed. T1c-T2a, T2b-T2c:Clinical tumor Stages at initial diagnosis; N0:Clinical lymph node stage at initial diagnosis; M0:Distant metastasis.
  Participants
    Low | 61 | 60 | 121
    Intermediate | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostate Cancer Progression
Description: Time to cancer prostate progression (pathological or therapeutic): time (in months) from date of randomization until the date of cancer progression (pathological or therapeutic). Pathological progression: increase in primary or secondary Gleason pattern by greater than or equal (>=) 1 or higher proportion of cancer positive cores (>=15 percent [%] increase). Therapeutic progression: earliest occurrence of primary therapy for prostate cancer (prostatectomy/radiation/focal therapy/systemic therapy). Medians and 95% CIs were calculated with the Kaplan-Meier (KM) method. Participants with no cancer progression at the time of study completion, discontinuation or death were censored at the last assessment date. Participants switching therapy during the study were censored at the time of the initial therapy switch, and participants discontinuing therapy were censored at the time of study discontinuation.
Time Frame: From the date of randomization until the date of the cancer progression (pathological or therapeutic) (up to study completion date, 28 Aug 2020; approximately 50 months)
Population: FAS population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Months | NA [36.14 to NA] — Median and upper limit were not achieved due to low number of events. | NA [24.67 to NA] — Median and upper limit were not achieved due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide vs Active Surveillance; Test type: Superiority; p = 0.016, Log Rank — P-value was from a 2-sided stratified log-rank test; Hazard Ratio (HR) = 0.542, 95% CI 2-sided [0.330 to 0.892] — HR, 95% CI for HR:based on a Cox regression model assuming proportional hazards with treatment, prostate cancer risk,type of biopsy,baseline variables(as age, race), time since prostate cancer diagnosis as fixed effects and random effect of site

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE: any untoward medical occurrence in a participant administered study drug or who underwent study procedures and did not necessarily had a causal relationship with treatment. An abnormality identified during a medical test: an AE only if the abnormality induced clinical signs or symptoms, required active intervention, required interruption, or discontinuation of study medication, or was clinically significant in the opinion of investigator. An AE: serious if it resulted in any of the following outcomes: Death, was life-threatening, Persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, Congenital anomaly, or birth defect, Inpatient hospitalization or prolongation of hospitalization, Other medically important event. Drug-related AEs: assessed by investigator as AEs whose relationship to study drugs could not be ruled out.
Time Frame: From date of first dose of enzalutamide or randomization until end of study (up to study completion date, 28 Aug 2020; approximately 50 months)
Population: The safety analysis set (SAF) consisted of all participants who enrolled in the study and were randomized to receive study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 112 | 113
Participants
  Serious Adverse Events (SAEs) | 19 | 10
  non-SAEs | 103 | 67

3. Secondary Outcome: Percentage of Participants Reported Negative Biopsies for Cancer
Description: Percentage of Participants who reported negative biopsies for cancer were reported.
Time Frame: At the end of months 12 and 24
Population: FAS population with available data at each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Percentage of participants
  At the end of month 12 | 35.1 | 14.2
  At the end of month 24: number analyzed (Participants) | 100 | 83
  At the end of month 24 | 19.0 | 12.0
Statistical Analysis 1: Comparison: Enzalutamide vs Active Surveillance; At the end of month 12; Test type: Superiority; p = 0.00, Regression, Logistic — P-value: Based on the exact binomial distribution from the logistic regression model; Odds Ratio (OR) = 3.5, 95% CI 2-sided [1.76 to 6.92] — OR: from logistic regression model where fixed covariates=treatment group, prostate cancer risk, type of biopsy, age, race and time since prostate cancer diagnosis; random effects: site and subject. 95% CI: based on exact binomial distribution
Statistical Analysis 2: Comparison: Enzalutamide vs Active Surveillance; At the end of month 24; Test type: Superiority; p = 0.289, Regression, Logistic — P-value: Based on the exact binomial distribution from the logistic regression model; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.66 to 4.00] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Percent of Cancer Positive Cores at Month 12 and 24
Description: Percent positive cores were calculated using the number of systemically sampled prostate regions and any targeted regions with at least 1 positive core divided by the total number of systematically sampled regions and targeted regions. This implied that despite the number of samples within a given systematic or targeted region, any positive core indicated that region as positive.
Time Frame: Baseline, months 12 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Percent of Cancer positive cores
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Percent of Cancer positive cores
  Change at month 12: number analyzed (Participants) | 90 | 81
  Change at month 12 | -14.2 (15.68) | -1.9 (14.70)
  Change at month 24: number analyzed (Participants) | 53 | 42
  Change at month 24 | -7.3 (17.74) | -0.8 (21.62)
Statistical Analysis 1: Comparison: Enzalutamide vs Active Surveillance; Change at month 12; Test type: Superiority; p < 0.001, Mixed Models Analysis — P-values: from differences of least squares means.Bonferroni-Holm was used in the primary hypothesis testing to adjust for multiplicity; Compound symmetry was used as the covariance structure. Covariance parameters:estimated using Restricted Maximum likelihood; LS mean difference = -10.07, 95% CI 2-sided [-14.79 to -5.34], Standard Error of Mean 2.398 — Mixed model repeated measure(MMRM) with treatment group, prostate cancer risk(low/intermediate), type of biopsy(mpMRI-targeted/non-mpMRI-targeted), visit, visit-by-treatment, baseline scores as fixed factors, site and participants as random factors
Statistical Analysis 2: Comparison: Enzalutamide vs Active Surveillance; Change at month 24; Test type: Superiority; p = 0.1063, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; LS mean difference = -5.15, 95% CI 2-sided [-11.40 to 1.11], Standard Error of Mean 3.174 — MMRM with treatment group, prostate cancer risk (low vs. intermediate), type of biopsy (mpMRI targeted vs. non mpMRI targeted), visit, visit-by-treatment and baseline scores were the fixed factors, and site and participants were the random factors

5. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as time in months from the date of randomization or first dose enzalutamide untill date of PSA progression (secondary rise in serum PSA >=25% above baseline or >=25% above nadir or absolute increase >= 2 nanogram per mililiter [ng/mL]). Participants with no PSA progression at the time of trial completion, discontinuation or death were censored at the last assessment date. Additionally, participants switching therapy during the study were censored at the time of the initial therapy switch, and participants discontinuing therapy were censored at the time of study discontinuation. Medians and 95% CIs were calculated with the KM method.
Time Frame: From date of randomization or first dose of enzalutamide until date of PSA progression (pathological or therapeutic) (up to study completion date=28 Aug 2020, median duration: 14.82 months for "Enzalutamide", 8.80 months for "Active Surveillance")
Population: FAS population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Months | 14.82 [14.75 to 14.95] | 8.80 [6.05 to 11.53]
Statistical Analysis 1: Comparison: Enzalutamide vs Active Surveillance; Test type: Superiority; p = 0.032, Log Rank — P-value: from a 2-sided, stratified log-rank test; Hazard Ratio (HR) = 0.714, 95% CI 2-sided [0.525 to 0.972] — HR and 95% CI for HR:based on Cox regression model assuming proportional hazards with treatment, prostate cancer risk, type of biopsy, baseline variables(as age, race), time since prostate cancer diagnosis as fixed effects and random effect of site

6. Secondary Outcome: Percentage of Participants With Secondary Rise in Serum PSA
Description: Percentage of participants with secondary rise in serum PSA > 25% baseline or > 25% above nadir or absolute increase >2 ng/mL were reported in this measure.
Time Frame: At the end of months 12, 24 and at the end of study (up to study completion date, 28 Aug 2020, approximately 50 months)
Population: FAS population with available data at each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Percentage of participants
  At the end of month 12 | 24.6 | 69.0
  At the end of month 24: number analyzed (Participants) | 100 | 83
  At the end of month 24 | 92.0 | 92.8
  At the end of study: number analyzed (Participants) | 69 | 52
  At the end of study | 100.0 | 96.2
Statistical Analysis 1: Comparison: Enzalutamide vs Active Surveillance; At the end of month 12; Test type: Superiority; p = 0.000, Regression, Logistic — P-value:based on the exact binomial distribution from the logistic regression model; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.08 to 0.26] — OR:from logistic regression model where treatment group, prostate cancer risk, type of biopsy, age, race and time since prostate cancer diagnosis were fixed covariates, site and participant were random effects. 95% CI:based on binomial distribution
Statistical Analysis 2: Comparison: Enzalutamide vs Active Surveillance; At the end of month 24; Test type: Superiority; p = 0.807, Regression, Logistic — P-value: based on the exact binomial distribution from the logistic regression model; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.37 to 3.53] — OR: from logistic regression model where treatment group, prostate cancer risk, type of biopsy, age, race and time since prostate cancer diagnosis were fixed covariates, site and participant were random effects. 95% CI:based on binomial distribution
Statistical Analysis 3: Comparison: Enzalutamide vs Active Surveillance; At the end of study; Test type: Superiority; p = 0.931, Regression, Logistic — P-value:based on the exact binomial distribution from the logistic regression model; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.50 to 2.15] — [estimate comment as in outcome 6, analysis 2]

7. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI) Questionnaire Composite Scores to Months 3, 6, 12, 18 and 24
Description: The BFI is a screening tool designed to assess the severity and impact of fatigue on daily functioning of participants with cancer during the 24 hours. There are 9 items on the scale. The first three questions ask participants to rate their fatigues on a scale from 0 (no fatigue) - 10 (as bad as you can imagine), with higher scores indicating worse outcome. The remaining six questions ask participants to rate how much fatigue has interfered with their daily activities on a scale from 0 (Does not interfere) to 10 (Completely interferes). A composite fatigue score was obtained by averaging all the items on the BFI, ranged between 0 to 10, with a higher BFI fatigue score indicating worse outcome. The composite BFI score was calculated only if at least 5 of the 9 items were answered.
Time Frame: Baseline, months 3, 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 3: number analyzed (Participants) | 102 | 106
  Change at month 3 | 0.7 (1.67) | 0.0 (1.32)
  Change at month 6: number analyzed (Participants) | 97 | 102
  Change at month 6 | 1.0 (2.03) | -0.1 (1.27)
  Change at month 12: number analyzed (Participants) | 93 | 87
  Change at month 12 | 1.2 (1.94) | 0.1 (1.32)
  Change at month 18: number analyzed (Participants) | 77 | 58
  Change at month 18 | 0.3 (1.43) | -0.2 (1.22)
  Change at month 24: number analyzed (Participants) | 68 | 46
  Change at month 24 | 0.5 (1.15) | 0.1 (1.27)

8. Secondary Outcome: Change From Baseline in 12-Item Short Form Survey (SF-12) Questionnaire Composite Score to Months 6, 12, 18, 24 - Mental Component Summary
Description: SF-12 is a questionnaire that measures overall health related quality of life using 12 questions. The questions are then scored and weighted into 2 subscales, physical health and mental health. Each yields scores from 0 (representing the worst possible debilitation) to 100 (representing no reduction in quality of life). Scores are transformed and ranges between 0 to 100; higher score indicates improvement.
Time Frame: Baseline, months 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 6: number analyzed (Participants) | 96 | 102
  Change at month 6 | -1.6 (5.94) | -0.1 (6.83)
  Change at month 12: number analyzed (Participants) | 93 | 88
  Change at month 12 | -2.3 (6.70) | -1.7 (6.84)
  Change at month 18: number analyzed (Participants) | 77 | 58
  Change at month 18 | 0.0 (6.18) | -0.5 (5.24)
  Change at month 24: number analyzed (Participants) | 67 | 46
  Change at month 24 | -0.3 (5.27) | -1.4 (7.29)

9. Secondary Outcome: Change From Baseline in SF-12 Questionnaire Composite Score to Months 6, 12, 18, 24 - Physical Component Summary
Description: as for outcome 8
Time Frame: Baseline, months 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 6: number analyzed (Participants) | 96 | 102
  Change at month 6 | -2.8 (6.64) | 0.1 (5.45)
  Change at month 12: number analyzed (Participants) | 93 | 88
  Change at month 12 | -3.9 (6.73) | -0.9 (5.52)
  Change at month 18: number analyzed (Participants) | 77 | 58
  Change at month 18 | -3.9 (6.37) | -0.4 (4.37)
  Change at month 24: number analyzed (Participants) | 67 | 46
  Change at month 24 | -2.8 (5.96) | -1.6 (5.42)

10. Secondary Outcome: Change From Baseline in The Expanded Prostate Cancer Index Composite (EPIC) Hormonal Assessment Scores at Months 6, 12, 18 and 24
Description: The EPIC Hormonal Assessment was a questionnaire used to measure quality of life (QoL) issues in participants with prostate cancer. There were a total of 6 questions related to hormonal function such as hot flashes, breast tenderness, depression, lack of energy, weight fluctuation. The answers ranged from "more than once a day" to "rarely or never" (ranged from 1 to 5, corresponding standardized scores were 100, 75, 50, 25, 0), "no problem" to "big problem" (ranged from 0 to 4, corresponding standardized scores were 100, 75, 50, 25, 0). Score from each answer was converted into standardized score at each visit. Total score was calculated by taking average of standardized scores. Total score was measured on a scale ranged from 0 (worst) to 100 (best) scale with higher scores representing better hormonal function.
Time Frame: Baseline, months 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 6: number analyzed (Participants) | 98 | 101
  Change at month 6 | 2.2 (6.74) | 0.2 (3.51)
  Change at month 12: number analyzed (Participants) | 93 | 87
  Change at month 12 | -1.1 (6.77) | 0.4 (4.45)
  Change at month 18: number analyzed (Participants) | 78 | 57
  Change at month 18 | -1.7 (3.81) | -0.5 (4.29)
  Change at month 24: number analyzed (Participants) | 68 | 45
  Change at month 24 | -1.2 (4.93) | 0.6 (3.92)

11. Secondary Outcome: Change From Baseline in EPIC Sexual Assessment Scores at Months 6, 12, 18 and 24
Description: EPIC Sexual Assessment: a questionnaire to measure QoL issues in participants with prostate cancer, included a total of 9 questions on sexual function as level of sexual desire, ability to have an erection, ability to reach orgasm, quality and frequency of erections, frequency of sexual intercourse. Answers ranged from "very poor" to "very good,"(ranged from 1 - 5, corresponding standardized scores:0, 25, 50, 75, 100), "none" to "enough"(ranged from 1 - 4, corresponding standardized scores:0, 33, 67, 100), "no problem" to "big problem"(ranged from 0 - 4, corresponding standardized scores:100, 75, 50, 25, 0), and "never" to "daily"(ranged from 1 - 5, corresponding standardized scores:100, 75, 50, 25, 0). Scores from each answer was converted into standardized score at each visit. Total score = calculated by taking average of standardized scores. Total score was measured on a scale ranged from 0 (worst) to 100 (best), higher scores = better sexual function and satisfaction.
Time Frame: Baseline, months 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 6: number analyzed (Participants) | 96 | 99
  Change at month 6 | -26.7 (21.91) | -2.3 (15.34)
  Change at month 12: number analyzed (Participants) | 92 | 85
  Change at month 12 | -30.5 (23.31) | -2.9 (15.59)
  Change at month 18: number analyzed (Participants) | 77 | 58
  Change at month 18 | -9.5 (17.41) | -2.1 (15.91)
  Change at month 24: number analyzed (Participants) | 67 | 46
  Change at month 24 | -12.2 (18.35) | -3.7 (16.81)

12. Secondary Outcome: Change From Baseline in EPIC Urinary Assessment Scores at Month 6, 12, 18 and 24
Description: EPIC urinary assessment: a questionnaire to measure QoL issues in participants with prostate cancer, included a total of 7 questions on urinary function as leaking urine, blood in urine, pain/burning on urination, urinary control and frequency. Answers ranged from "more than once a day" to "rarely or never"(scores from 1 - 5,corresponding standardized scores[CSS]:0, 25, 50, 75, 100), "no urinary control" to "full urinary control"(scores from 1 - 4,CSS:0, 33, 67, 100), "none" to "3 or more pads per day"(scores from 0 - 3, CSS:100, 67, 33, 0), "no problem" to "big problem"(scores from 0 - 4, CSS:100, 75, 50, 25, 0), and "no problem" to "big problem"(scores from 1 - 5, corresponding standardized score:100, 75, 50, 25, 0). Score from each answer was converted into a corresponding standardized score at each visit. Total score was calculated by taking average of standardized scores. Total score ranged from 0(worst) to 100(best), higher scores = better urinary function.
Time Frame: Baseline, months 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 6: number analyzed (Participants) | 97 | 102
  Change at month 6 | -2.7 (10.26) | 0.7 (10.28)
  Change at month 12: number analyzed (Participants) | 94 | 86
  Change at month 12 | -4.2 (10.10) | 0.3 (10.98)
  Change at month 18: number analyzed (Participants) | 78 | 56
  Change at month 18 | -1.6 (9.55) | 0.2 (12.91)
  Change at month 24: number analyzed (Participants) | 69 | 45
  Change at month 24 | -1.6 (9.36) | 0.3 (13.47)

13. Secondary Outcome: Change From Baseline in Memorial Anxiety Scale for Prostate Cancer (MAX-PC) Scores at Months 6, 12, 18 and 24
Description: The MAX-PC was a questionnaire used to assess participants' feelings about prostate cancer and PSA tests. There were a total of 18 questions related to understanding how participants cope with aspects of their treatment and medical tests frequently involved in their care; questions such as strong feelings about prostate cancer, scared of PSA tests, trouble sleeping due to thoughts of prostate cancer, unable to plan for the future due to prostate cancer, fear of cancer getting worse. The answers range from "not at all" to "often" and "strongly disagree" to "strongly agree. Total score ranged from 0-54, an increase in the score indicates a worsened anxiety level.
Time Frame: Baseline, months 6, 12, 18 and 24
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enzalutamide | Active Surveillance
Number analyzed (Participants) | 114 | 113
Units on a scale
  Change at month 6: number analyzed (Participants) | 96 | 102
  Change at month 6 | -1.6 (6.23) | -0.5 (4.45)
  Change at month 12: number analyzed (Participants) | 92 | 88
  Change at month 12 | -0.8 (4.49) | -0.0 (4.52)
  Change at month 18: number analyzed (Participants) | 77 | 58
  Change at month 18 | -1.3 (4.86) | -0.6 (4.70)
  Change at month 24: number analyzed (Participants) | 68 | 46
  Change at month 24 | -1.4 (5.19) | -0.6 (3.78)

ADVERSE EVENTS:
Time Frame: From date of first dose of enzalutamide or randomization until end of study (up to study completion date, 28 Aug 2020, approximately 50 months)
Arm/Group | Enzalutamide | Active Surveillance
All-Cause Mortality (participants affected / at risk) | 3/112 | 0/113
Serious Adverse Events (participants affected / at risk) | 19/112 | 10/113
Other Adverse Events (participants affected / at risk) | 101/112 | 34/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=112) | Active Surveillance (N=113)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Central cord syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electroencephalogram abnormal (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Physical disability (Social circumstances) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=112) | Active Surveillance (N=113)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (1)
Fatigue (General disorders) | 62 (68) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 6 (6)
Weight decreased (Investigations) | 6 (6) | 2 (2)
Weight increased (Investigations) | 6 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Libido decreased (Psychiatric disorders) | 10 (10) | 1 (1)
Dysuria (Renal and urinary disorders) | 6 (6) | 5 (7)
Pollakiuria (Renal and urinary disorders) | 8 (8) | 4 (4)
Breast enlargement (Reproductive system and breast disorders) | 7 (8) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 29 (31) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 22 (22) | 4 (4)
Gynaecomastia (Reproductive system and breast disorders) | 42 (45) | 3 (3)
Nipple pain (Reproductive system and breast disorders) | 34 (34) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0)
Hot flush (Vascular disorders) | 6 (6) | 0 (0)
Hypertension (Vascular disorders) | 10 (11) | 10 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02799745/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT02799745/SAP_001.pdf